CLINICAL TRIAL: NCT03497221
Title: Simulation and Visual Identity as a Patient Safety Strategy in the Care of Nasoenteric Tube: Clinical Trial
Brief Title: Education Intervention as a Patient Safety Strategy in the Care of Nasoenteric Tube
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 63247916500005327
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Patient Safety; Enteral Nutrition
Keywords: Nursing Education
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education intervention (Other): The educational intervention is based on a hospital institutional protocol for patient using enteral tubes. A clinical simulation will be performed using a low fidelity manikin, where nursing technicians will identify and correct erros, such as: inconsistency between the patient's identification and the diet label, the administration of the diet with a low headboard, fixation of tube not detached and dirty, delay of the diet and others. The simulation will be described through a guide.
  Interventions: Behavioral: Education intervention
- Visual identity campaign (Other): The visual identity will be given by a set of actions, called "campaign". The campaign consists in the creation and implantation of different materials to be used at the bedside of the patients in use of diet by SNE, such as: (a) poster summarizing care, (b) colored adhesive label to identify devices (c) badge with safety care reminders.
  Interventions: Behavioral: Visual identity campaign

INTERVENTIONS:
Behavioral: Education intervention — The same description of arm Education intervention.
  Arms: Education intervention
Behavioral: Visual identity campaign — The same description of arm Visual identity campaign.
  Arms: Visual identity campaign

SUMMARY:
The safety of the patient using a nasoenteral tube depends on the constant evaluation of the nursing team. The most implemented strategies for safe practice are education interventions, however, seem insufficient to change behavior. Active methodologies may be more promising alternatives for the development of these competencies. The objective is evaluate the effect of an isolated education intervention and combined with a visual identity campaign on the safe practice in the use of nursing care to the patient in use nasoenteral tubes. The clinical trial will be carried out in 2017, in a university hospital. Two profiles of participants will be included in the study: the first one refers to the nursing technicians of the hospital areas, part of them will receive a set of interventions, and the second one refers to the patients in use nasoenteral tube, considering that the effect of intervention will be measured by assessing compliance with care routines.

DETAILED DESCRIPTION:
The safety of the patient undergoing enteral nutritional therapy depends on the constant evaluation of the nursing team, which, through specific skills, allows the establishment of nutritional care and prevents incidents related to the diet administration process. The challenge is to adopt safe practices that contemplate all these specificities, knowing that only knowledge is insufficient for the development of these competences, but also depends on the ability and commitment of these professionals.

Training and capacity are predominant strategies in the health area to increase patient safety in the execution of nursing staff's care activities, however, this type of approach, when applied in isolation, is sometimes insufficient to change behavior end development of skills and attitudes among these professionals. Combined strategies such as alerts and reminders systems, educational visits, auditing systems, clinical simulations, feedbacks and workshops, on clinical practice safety are being deployed and evaluated as a more effective way of changing behavior.

In this sense, the research question of the present project is: The implementation of a strategy of safety in service through an educational intervention associated to the visual identity campaign is able to increase the adhesion of the nursing technicians to the fulfillment of routines in the use of nasoenteral tube? The objective is evaluate the effect of an isolated education intervention and combined with a visual identity campaign on the safe practice in the use of nursing care to the patient in use nasoenteral tubes. The clinical trial will be carried out in 2017, in a university hospital. Two profiles of participants will be included in the study: the first one refers to the nursing technicians of the hospital areas, part of them will receive a set of interventions, and the second one refers to the patients in use nasoenteral tube, considering that the effect of intervention will be measured by assessing compliance with care routines.

The study will be conducted according to the following steps, respectively: (1) Evaluation of the agreement between observers, (2) Pre-intervention evaluation (baseline), (3) Intervention (Educational Intervention and Visual Identity Campaign) and (4) Post-intervention evaluation. Both groups (IG and CG) will be submitted to the same research procedures in the evaluation stages (pre- and post-intervention); However, only the nursing technicians of the GI will be submitted to an intervention stage.

ELIGIBILITY:
Inclusion Criteria:

* Nursing technicians: All nursing technicians of the intervention units will be potentially eligible for the study.
* Patients: with nasoenteral tube, adults (18 years of age or older) and who are hospitalized in the IG or CG units.

Exclusion Criteria:

* Workers who are not working during data collection. The nursing technicians who are part of the IG will be that could be reassigned to one of the units of the CG and vice versa.
* Patient: unaccompanied patients who are confused and / or disoriented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1084 (Estimated)
Dates: Start 2017-06-03 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Absence of conformity of nursing care in enteral nutritional therapy (ENT) with recommendations of good practices according to institutional protocols. | 12 months
  This outcome have been measured by means of a Nasoenteric Tube (NT) care checklist observed at the patient's bedside. The checklist contains 25 items that evaluate: Conference of labels and validity of the diets and water bottles and devices used for administration at NT; observation of head of bed routines during enteral infusions, correct NT fixation, hygiene of devices and infusion pumps used ENT.

SECONDARY OUTCOMES:
The presence of adverse event related to obstruction NT | 12 months
  This outcome have been measured through the evaluation of the records of the professional health team (nurses, doctors, nutritionists and nursing technicians).
The presence of adverse event related to displacement NT non-programmed | 12 months
  This outcome have been measured through the evaluation of the records of the professional health team (nurses, doctors, nutritionists and nursing technicians).
The presence of adverse event related to withdrawal NT non-programmed | 12 months
  This outcome have been measured through the evaluation of the records of the professional health team (nurses, doctors, nutritionists and nursing technicians).
The presence of adverse event related to administration of enteral diet by probe not positioned in the gastrointestinal tract | 12 months
  This outcome have been measured through the evaluation of the records of the professional health team (nurses, doctors, nutritionists and nursing technicians).
The presence of adverse event related to non-administration of enteral diet (partial or full) when suspension was not planned | 12 months
  This outcome have been measured through the evaluation of the records of the professional health team (nurses, doctors, nutritionists and nursing technicians).
The presence of adverse event related to cases of diarrhea (three or more episodes of soft or liquid stools within 24 hours) | 12 months
  This outcome have been measured through the evaluation of the records of the professional health team (nurses, doctors, nutritionists and nursing technicians).
The presence of adverse event related to cases of constipation (a disorder characterized by persistent difficulty of evacuation or a sensation of incomplete evacuation and / or infrequent bowel movements for at least 3 days) | 12 months
  This outcome have been measured through the evaluation of the records of the professional health team (nurses, doctors, nutritionists and nursing technicians).

CONTACTS AND LOCATIONS:
Overall Officials: Mariur G Beghetto, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided